CLINICAL TRIAL: NCT01729728
Title: Open-label Evaluation of the Pharmacokinetic Profile, Safety, and Efficacy of Tapentadol Oral Solution for the Treatment of Post-surgical Pain in Children and Adolescents Aged From 2 Years to Less Than 18 Years.
Brief Title: Pharmacokinetic, Efficacy and Safety Study of Tapentadol Oral Solution in Children With Postoperative Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Grünenthal GmbH (Industry)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KF5503/68; 2013-002016-27 (EudraCT Number)
Record Dates: First submitted 2012-11-06; First posted 2012-11-20 (Estimated); Results first posted 2014-11-27 (Estimated); Last update posted 2019-11-04 (Actual); Status verified 2019-10

CONDITIONS: Postoperative Pain; Acute Pain
Keywords: Tonsillectomy; Dental surgery; Ear surgery; Nose surgery; Throat surgery
MeSH Terms: conditions — Pain, Postoperative; Acute Pain | interventions — Tapentadol

ARMS (1):
- Tapentadol (Experimental)
  Interventions: Drug: Tapentadol

INTERVENTIONS:
Drug: Tapentadol — Tapentadol oral solution single dose (1mg/kg body weight)

SUMMARY:
To find out if a drug called tapentadol administered by mouth safely relieves pain in children. Look at the amount of tapentadol in the blood after a single oral dose.

Tapentadol oral solution for children is still being tested and is not yet registered. Tapentadol tablets are effective in treating both acute and chronic pain in adults. This trial will help to understand how tapentadol oral solution works in children.

DETAILED DESCRIPTION:
The lower age limit for the clinical trial was initially set to 3 years of age in the protocol. The trial planned for the inclusion of participants in three age categories. Age 3 to less than 6 years (young children), age 6 to less than 12 years (older children) and age 12 to less than 18 years of age (adolescents). There was a request by the Paediatric Committee (PDCO) at the European Medicines Agency to include participants 2 years of age (very young children). The protocol amendment thus planned to combine the two youngest age groups into a single reporting group. The protocol amendment only planned that the very young children group would have separate analysis for the Faces Pain Scale Revised (FPS-R) Scale and for the presentation of the serum concentrations, because the pharmacokinetic sampling scheme used in the 2 year old participants was different from the young children group (aged 3 to less than 6 years).

ELIGIBILITY:
Inclusion Criteria:

* A maximum body weight of 85.0 kg.
* A minimum body weight of 10 kg for participants aged 2 years to less than 3 years old.
* If female and post-menarchal, or 12 years or older, the subject has a negative urine pregnancy test within 24 hours before surgery.
* Having completed either dental surgery or tonsillectomy with or without adenoidectomy surgery (age group: 6 to less than 18 years of age).
* Having completed ear, nose, or throat surgery (including but not limited to tonsillectomy (age group: 2 to less than 3 years of age).
* Participant aged 6 to less than 18 years has a post-operative pain intensity score greater than or equal to 4 on the Color Analog Scale (CAS) as a result of the surgical procedure or the participant has a pain level that the usual standard of care following the surgical procedure (which reliably produces moderate to severe pain) requires opioid treatment.
* Participant aged 2 years to less than 6 years has a pain level following a surgical procedure that reliably produces moderate to severe pain, for which the usual standard of care requires opioid treatment.
* Participant is alert, orientated, and able to follow commands and complete the post-operative required procedures.

Exclusion Criteria:

* History of brain injury.
* Clinically relevant abnormal ECG.
* Clinically unstable vital signs and/or a saturation of oxygen saturation (SpO2) less than 93%. During surgery SpO2 may decrease <93%.
* Clinically relevant abnormal values for clinical chemistry, hematology, or urinalysis at enrollment.
* Body temperature above 38.5°C within 48 hours prior to dosing.
* Positive drugs of abuse test result.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 86 (Actual)
Dates: Start 2012-11; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Grünenthal GmbH
Locations (1):
- Jean Brown Research, Salt Lake City, Utah, United States

REFERENCES:
- [Result] Muse D, Tarau E, Lefeber C, Sohns M, Brett M, Goldberg J, Rosenburg R. Pharmacokinetics, safety, and efficacy of tapentadol oral solution for treating moderate to severe pain in pediatric patients. J Pain Res. 2019 May 31;12:1777-1790. doi: 10.2147/JPR.S197039. eCollection 2019. PMID 31213888

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first participant was enrolled on the 15 Nov 2012 and the last participant completed the trial on the 24 Feb 2014.
Pre-assignment Details: Consent was obtained for 86 participants in the trial. 66 participants were allocated and received study drug (investigational medicinal product). Pharmacokinetic data was obtained for the planned 56 participants.
Groups:
- Adolescents: Single Dose of Tapentadol Oral Solution in Adolescents Age 12 to Less Than 18 Years. Tapentadol oral solution single dose (1mg/kg body weight)
- Older Children: Single Dose of Tapentadol Oral Solution in Children Age 6 to Less Than 12 Years. Tapentadol oral solution single dose (1mg/kg body weight)
- Young and Very Young Children: Single Dose of Tapentadol Oral Solution in Children Age 2 to Less Than 6 Years. Tapentadol oral solution single dose (1mg/kg body weight)
Period: Overall Study
Arm/Group | Adolescents | Older Children | Young and Very Young Children
Started | 21 | 28 | 17
Completed | 20 | 22 | 16
Not Completed | 1 | 6 | 1
Not completed — Adverse Event | 0 | 6 | 0
Not completed — Protocol Violation | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Number of participants that were dosed.
Groups:
- Total: Total of all reporting groups
Arm/Group | Adolescents | Older Children | Young and Very Young Children | Total
Number analyzed (Participants) | 21 | 28 | 17 | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.5 (1.6) | 8.3 (1.6) | 3.4 (1.1) | 9.3 (4.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 17 | 8 | 34
  Male | 12 | 11 | 9 | 32
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1
  White | 21 | 27 | 15 | 63
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 21 | 28 | 17 | 66
Weight [Mean (Standard Deviation); unit: kilograms] | 61.30 (9.78) | 28.85 (5.89) | 16.34 (2.20) | 35.95 (19.36)
Height [Mean (Standard Deviation); unit: centimeter] | 170.6 (10.7) | 132.9 (11.1) | 101.7 (8.1) | 136.9 (28.3)

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetic Profile of Serum Concentrations of Tapentadol After a Single Dose of Tapentadol Oral Solution in Adolescents (Age 12 to Less Than 18 Years).
Description: Mean and Standard Deviation of Serum Concentrations of Tapentadol. Serum was analyzed by means of liquid chromatography coupled to tandem mass spectrometry with a lower limit of quantification (LLOQ) at 0.2 ng/mL.
Time Frame: up to 15 hours
Population: Pharmacokinetic Set
Measure: Mean (Standard Deviation); unit: nanogram per milliliter
Groups:
- Tapentadol Serum Concentrations: Adolescents: Tapentadol oral solution single dose (1mg/kg body weight). Participants aged 12 years and less than 18 years of age.
Arm/Group | Tapentadol Serum Concentrations: Adolescents
Number analyzed (Participants) | 19
nanogram per milliliter
  15 minutes post-dose | 23.2 (34.0)
  30 minutes post-dose: number analyzed (Participants) | 18
  30 minutes post-dose | 45.6 (33.0)
  1 hour post-dose: number analyzed (Participants) | 18
  1 hour post-dose | 49.4 (21.2)
  2 hours post-dose: number analyzed (Participants) | 18
  2 hours post-dose | 43.1 (14.2)
  4 hours post-dose: number analyzed (Participants) | 17
  4 hours post-dose | 32.8 (10.8)
  6 hours post-dose: number analyzed (Participants) | 18
  6 hours post-dose | 22.3 (11.9)
  11 hours post-dose: number analyzed (Participants) | 18
  11 hours post-dose | 8.14 (6.35)
  15 hours post-dose: number analyzed (Participants) | 17
  15 hours post-dose | 3.66 (3.26)

2. Secondary Outcome: Pain Intensity Assessments Using the Visual Analog Scale (VAS) in Adolescents (Age 12 to Less Than 18 Years).
Description: At predefined times after investigational medicinal product administration, participants were asked to rate their pain on a 100 mm line (visual analog scale - VAS) by marking a point on the line in response to:
  "My pain at this time is". The mark was scored between "no pain" and " pain as bad as it could be". The distance was then measured by a clinician and reported.
  A value of 0 indicates "no pain". A value of 100 indicates "pain as bad as it could be".
Time Frame: Baseline; 15 hours
Population: Protocol pre-specified reporting groups.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Visual Analog Scale: Adolescents: Single Dose of Tapentadol Oral Solution in Adolescents Age 12 to Less Than 18 Years. Tapentadol oral solution single dose (1mg/kg body weight).
Arm/Group | Visual Analog Scale: Adolescents
Number analyzed (Participants) | 21
units on a scale
  Pre-dose | 71.5 (13.3)
  15 minutes post-dose | 63.6 (24.4)
  30 minutes post-dose | 53.2 (27.3)
  1 hour post-dose | 46.3 (26.5)
  2 hours post-dose: number analyzed (Participants) | 20
  2 hours post-dose | 34.0 (24.6)
  4 hours post-dose: number analyzed (Participants) | 20
  4 hours post-dose | 43.5 (26.8)
  6 hours post-dose: number analyzed (Participants) | 20
  6 hours post-dose | 34.8 (24.3)
  11 hours post-dose: number analyzed (Participants) | 20
  11 hours post-dose | 32.7 (21.1)
  15 hours post-dose: number analyzed (Participants) | 20
  15 hours post-dose | 33.4 (20.1)

3. Secondary Outcome: Pain Intensity Assessments Using the McGrath Color Analog Scale in Adolescent Participants and Older Children (Age 6 to Less Than 18 Years).
Description: Pain intensity assessments were with a 0 (no pain) to 10 (worst pain) scored McGrath color analog scale (CAS) in participants aged 6 years to less than 18 years, i.e. in Adolescents and Older Children. Participants were presented with the CAS and instructed to place the sliding bar on the color that best represented their pain intensity level at the time of assessment. The CAS is a pocket size tool used to measure the self-reported pain intensity of the older participants. The CAS consists of a 145 mm long triangular shaped strip of plastic, varying in width and hue from 1 mm wide and light pink hue at the bottom (and text no pain), to 3 mm wide and deep red hue at the top (most pain). This instrument includes 2 sides. One side shows the color pain intensity scale as described and the other shows a graduated scale, which provides a specific numeric value for the participant-reported level of pain.
Time Frame: Baseline; 15 hours post-dose
Population: Protocol pre-specified reporting groups.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- McGrath Color Analog Scale: Adolescents: Single Dose of Tapentadol Oral Solution in Adolescents Age 12 to Less Than 18 Years. Tapentadol oral solution single dose (1mg/kg body weight).
- McGrath Color Analog Scale: Older Children: Single Dose of Tapentadol Oral Solution in Children Age 6 to Less Than 12 Years. Tapentadol oral solution single dose (1mg/kg body weight).
Arm/Group | McGrath Color Analog Scale: Adolescents | McGrath Color Analog Scale: Older Children
Number analyzed (Participants) | 21 | 28
units on a scale
  Pre-dose | 6.643 (1.461) | 4.670 (1.602)
  15 minutes post-dose | 6.131 (2.180) | 3.071 (1.718)
  30 minutes after dosing | 5.262 (2.311) | 2.571 (1.824)
  1 hour post-dose | 4.393 (2.299) | 2.407 (1.723)
  2 hours post-dose | 3.475 (2.173) | 2.292 (1.793)
  4 hours post-dose | 4.200 (2.113) | 2.341 (1.899)
  6 hours post-dose | 3.438 (1.960) | 2.636 (2.152)
  11 hours post-dose | 3.350 (1.836) | 3.352 (1.851)
  15 hours post-dose | 3.288 (1.578) | 3.568 (2.549)

4. Secondary Outcome: Pain Intensity Assessments Using the Faces Pain Scale (Revised) in Children Age 3 to Less Than 12 Years.
Description: This assessment tool was used in 3 to less than 12 year old participants, i.e. Older Children and Young Children.
  The Faces Pain Scale (Revised) [FPS-R] score as allocated to a selected face by the participant. There are 6 faces and the participant is asked to indicate on a face to express how much it hurts.
  The numeric value 0 (no pain) to 10 (very much pain) is read off the reverse side of the scale by the clinician.
Time Frame: Baseline; 15 hours post-dose
Population: The protocol pre-specified that the Faces Pain Scale (Revised) would not be administered in the very young participants (aged 2 to less than 3 years).
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Faces Pain Scale: Older Children: Single Dose of Tapentadol Oral Solution in Children Age 6 to Less Than 12 Years. Tapentadol oral solution single dose (1mg/kg body weight)
- Faces Pain Scale: Young Children: Single Dose of Tapentadol Oral Solution in Children Age 3 to Less Than 6 Years. Tapentadol oral solution single dose (1mg/kg body weight). The children aged 2 were assessed using the FLACC (Face, Legs, Activity, Cry, Consolability) Scale and not the 6-point Faces Pain Scale - Revised.
Arm/Group | Faces Pain Scale: Older Children | Faces Pain Scale: Young Children
Number analyzed (Participants) | 28 | 12
units on a scale
  Pre-dose | 4.8 (1.6) | 6.8 (3.2)
  15 minutes post-dose | 3.5 (1.8) | 4.5 (4.0)
  30 minutes post-dose | 2.9 (1.8) | 2.8 (3.2)
  1 hour post-dose | 2.4 (1.6) | 1.8 (3.3)
  2 hours post-dose | 2.6 (1.7) | 1.2 (2.9)
  4 hours post-dose | 2.5 (1.6) | 3.5 (3.2)
  6 hours post-dose | 2.7 (2.1) | 1.8 (2.3)
  11 hours post-dose | 2.7 (1.7) | 2.3 (2.4)
  15 hours post-dose | 3.5 (2.2) | 2.8 (2.9)

5. Secondary Outcome: Pain Intensity Assessment Using the Face, Legs, Activity, Cry, Consolability Scale in Young and Very Young Children (Age 2 to Less Than 6 Years).
Description: The Face Legs Activity Cry Consolability (FLACC) Scale was developed by the Department of Anesthesiology, University of Michigan Medical School and Health Systems. The FLACC Scale is a behavioral scale for scoring postoperative pain in children between the ages of two months and seven years or in persons unable to communicate. In this trial the scale was used in the young and very young children, i.e. in participants aged 2 to less than 6 years. This tool includes five categories of pain behaviors, including facial expression, leg movement, activity, cry, and consolability. The clinician observes the participant for 5 minutes or more and scores each category with a 0, 1 or 2. The scores are added together for a total score ranging from 0 (no pain) to 10 (worst pain). The higher the total score the higher the pain.
Time Frame: Baseline; 15 hours post-dose
Population: The protocol pre-specified that the young and very young children will be reported as one group.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Face, Legs, Activity, Cry, Consolability Scale: Single Dose of Tapentadol Oral Solution in Children Age 2 to Less Than 6 Years. Tapentadol oral solution single dose (1mg/kg body weight).
Arm/Group | Face, Legs, Activity, Cry, Consolability Scale
Number analyzed (Participants) | 17
units on a scale
  Pre-dose | 4.2 (2.2)
  15 minutes post-dose | 1.8 (1.6)
  30 minutes post-dose | 1.2 (1.6)
  1 hour post-dose | 1.1 (1.4)
  2 hours post-dose | 0.8 (1.1)
  4 hours post-dose | 1.5 (1.7)
  6 hours post-dose | 0.8 (1.6)
  11 hours post-dose | 0.9 (2.1)
  15 hours post-dose | 0.8 (1.2)

6. Secondary Outcome: Sum of Pain Intensity Differences Over the 4 Hours After Dosing Derived From the Different Pain Scales and for All Age Groups
Description: Different pain intensity assessment tools were used in the different age groups. Therefore the sum of pain intensities were calculated and are reported for each age group based on the tool used.
  Adolescents - Age 12 to Less Than 18 Years.
  Older Children - Age 6 to Less Than 12 Years.
  Young Children - Age 3 to Less Than 6 Years.
  Very Young Children - Age 2 to Less Than 3 Years.
  * CAS (McGrath color analog scale) [Theoretical Range: -40 to + 40],
  * VAS (100 mm Visual Analog Scale) [Theoretical Range: -400 to + 400],
  * FPS-R (6-point Faces Pain Scale - Revised) [Theoretical Range: -40 to + 40],
  * FLACC (Face, Legs, Activity, Cry, and Consolability score) [Theoretical Range: -40 to + 40].
  A mean score of zero indicates that there was no pain intensity change over the 4 hours.
  The positive values indicate that in the group as a whole the sum of all pain intensity values over the first 4 hours lead to a reduction in pain in the time period.
Time Frame: Baseline; 4 hours post-dose
Population: Protocol pre-specified reporting groups.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Sum of Pain Intensity Differences: The sum of pain intensity difference over 4 hours (SPID4) were calculated as the weighted sum of the scheduled pain intensity difference collected up to 4 hours after tapentadol oral solution administration.
  The time elapsed (in hours) since the previous measurement is multiplied with the pain intensity difference (PID) at the respective time, and defines the weight in the calculation of the weighted sum of pain intensity differences.
Arm/Group | Sum of Pain Intensity Differences
Number analyzed (Participants) | 65
units on a scale
  Adolescents SPID for VAS: number analyzed (Participants) | 20
  Adolescents SPID for VAS | 106.282 (75.350)
  Adolescents SPID for CAS: number analyzed (Participants) | 20
  Adolescents SPID for CAS | 8.925 (6.347)
  Older Children SPID for CAS: number analyzed (Participants) | 22
  Older Children SPID for CAS | 9.698 (7.610)
  Older Children SPID for FPS-R: number analyzed (Participants) | 22
  Older Children SPID for FPS-R | 8.724 (6.868)
  Young Children SPID for FPS-R: number analyzed (Participants) | 11
  Young Children SPID for FPS-R | 17.646 (14.674)
  Young Children SPID for FLACC: number analyzed (Participants) | 12
  Young Children SPID for FLACC | 11.614 (8.334)
  Very Young Children SPID for FLACC: number analyzed (Participants) | 4
  Very Young Children SPID for FLACC | 12.483 (8.955)

7. Primary Outcome: Pharmacokinetic Profile of Serum Concentrations of Tapentadol-O-glucuronide After a Single Dose of Tapentadol Oral Solution in Adolescents (Age 12 to Less Than 18 Years).
Description: Mean and Standard Deviation of Serum Concentrations of Tapentadol-O-glucuronide. Tapentadol-O-glucuronide is the metabolite of tapentadol. Metabolites are sometimes referred to as "breakdown products". The body alters the administered medication to a metabolite so that it can be more easily or quickly removed from the body. Tapentadol-O-glucuronide concentrations were measured in participants. Serum was analyzed by means of liquid chromatography coupled to tandem mass spectrometry with a lower limit of quantification (LLOQ) at 10 ng/mL.
Time Frame: up to 15 hours
Population: Pharmacokinetic Set
Measure: Mean (Standard Deviation); unit: nanogram per milliliter
Groups:
- Tapentadol-O-glucuronide Serum Concentrations: Adolescents: Tapentadol oral solution single dose (1mg/kg body weight). Participants aged 12 years and less than 18 years of age.
Arm/Group | Tapentadol-O-glucuronide Serum Concentrations: Adolescents
Number analyzed (Participants) | 18
nanogram per milliliter
  15 minutes post-dose | 404 (581)
  30 minutes post-dose: number analyzed (Participants) | 17
  30 minutes post-dose | 855 (672)
  1 hour post-dose: number analyzed (Participants) | 17
  1 hour post-dose | 1424 (542)
  2 hours post-dose | 1202 (366)
  4 hours post-dose: number analyzed (Participants) | 17
  4 hours post-dose | 824 (191)
  6 hours post-dose | 497 (138)
  11 hours post-dose | 150 (69.0)
  15 hours post-dose: number analyzed (Participants) | 17
  15 hours post-dose | 66.9 (35.4)

8. Primary Outcome: Pharmacokinetic Profile of Serum Concentrations of Tapentadol After a Single Dose of Tapentadol Oral Solution in Older Children (Age 6 to Less Than 12 Years).
Description: as for outcome 1
Time Frame: up to 15 hours
Measure: Mean (Standard Deviation); unit: nanogram per milliliter
Groups:
- Tapentadol Serum Concentrations: Older Children: Tapentadol oral solution single dose (1mg/kg body weight). Participants aged 6 years and less than 12 years of age.
Arm/Group | Tapentadol Serum Concentrations: Older Children
Number analyzed (Participants) | 22
nanogram per milliliter
  15 minutes to 1 hour post-dose (N=22) | 36.5 (21.8)
  1 to 4 hours post-dose (N=22) | 36.5 (15.7)
  4 to 11 hours post-dose (N=22) | 13.5 (6.52)
  11 to 15 hours post-dose (N=22) | 3.71 (1.96)

9. Primary Outcome: Pharmacokinetic Profile of Serum Concentrations of Tapentadol-O-glucuronide After a Single Dose of Tapentadol Oral Solution in Older Children (Age 6 to Less Than 12 Years).
Description: as for outcome 7
Time Frame: up to 15 hours
Population: Pharmacokinetic Set
Measure: Mean (Standard Deviation); unit: nanogram per milliliter
Groups:
- Tapentadol-O-glucuronide Serum Concentrations: Older Children: Tapentadol oral solution single dose (1mg/kg body weight). Participants aged 6 years and less than 12 years of age.
Arm/Group | Tapentadol-O-glucuronide Serum Concentrations: Older Children
Number analyzed (Participants) | 22
nanogram per milliliter
  15 minutes to 1 hour post-dose: number analyzed (Participants) | 20
  15 minutes to 1 hour post-dose | 676 (343)
  1 to 4 hours post-dose | 900 (330)
  4 to 11 hours post-dose | 321 (123)
  11 to 15 hours post-dose | 86.3 (37.8)

10. Primary Outcome: Pharmacokinetic Profile of Serum Concentrations of Tapentadol After a Single Dose of Tapentadol Oral Solution in Younger Children (Age 3 to Less Than 6 Years).
Description: as for outcome 1
Time Frame: up to 15 hours
Measure: Mean (Standard Deviation); unit: nanogram per milliliter
Groups:
- Tapentadol Serum Concentrations: Younger Children: Tapentadol oral solution single dose (1mg/kg body weight). Participants aged 3 years and less than 6 years of age.
Arm/Group | Tapentadol Serum Concentrations: Younger Children
Number analyzed (Participants) | 11
nanogram per milliliter
  15 minutes to 1 hour post-dose (N = 11) | 30.1 (19.2)
  4 to 11 hours post-dose (N=11) | 26.4 (10.7)

11. Primary Outcome: Pharmacokinetic Profile of Serum Concentrations of Tapentadol-O-glucuronide After a Single Dose of Tapentadol Oral Solution in Younger Children (Age 3 to Less Than 6 Years).
Description: as for outcome 7
Time Frame: up to 15 hours
Population: Pharmacokinetic Set
Measure: Mean (Standard Deviation); unit: nanogram per milliliter
Groups:
- Tapentadol-O-glucuronide Serum Concentrations Younger Children: Tapentadol oral solution single dose (1mg/kg body weight). Participants aged 3 years and less than 6 years of age.
Arm/Group | Tapentadol-O-glucuronide Serum Concentrations Younger Children
Number analyzed (Participants) | 11
nanogram per milliliter
  15 minutes to 1 hour post-dose: number analyzed (Participants) | 10
  15 minutes to 1 hour post-dose | 494 (377)
  4 to 11 hours post-dose | 504 (112)

12. Primary Outcome: Pharmacokinetic Profile of Serum Concentrations of Tapentadol After a Single Dose of Tapentadol Oral Solution in Very Young Children (Age 2 to Less Than 3 Years).
Description: as for outcome 1
Time Frame: up to 15 hours
Population: Pharmacokinetic Set
Measure: Mean (Standard Deviation); unit: nanogram per milliliter
Groups:
- Tapentadol Serum Concentrations: Very Young Children: Tapentadol oral solution single dose (1mg/kg body weight). Participants aged 2 years and less than 3 years of age.
Arm/Group | Tapentadol Serum Concentrations: Very Young Children
Number analyzed (Participants) | 4
nanogram per milliliter
  1.25 hours post-dose | 19.9 (13.2)
  3 hours post-dose | 37.7 (18.2)
  5 hours post-dose: number analyzed (Participants) | 3
  5 hours post-dose | 23.4 (6.36)
  8 hours post-dose | 10.0 (4.33)

13. Primary Outcome: Pharmacokinetic Profile of Serum Concentrations of Tapentadol-O-glucuronide After a Single Dose of Tapentadol Oral Solution in Very Young Children (Age 2 to Less Than 3 Years).
Description: as for outcome 7
Time Frame: up to 15 hours
Population: Pharmacokinetic Set
Measure: Mean (Standard Deviation); unit: nanogram per milliliter
Groups:
- Tapentadol-O-glucuronide Concentrations: Very Young Children: Tapentadol oral solution single dose (1mg/kg body weight). Participants aged 2 years and less than 3 years of age.
Arm/Group | Tapentadol-O-glucuronide Concentrations: Very Young Children
Number analyzed (Participants) | 4
nanogram per milliliter
  1.25 hours after administration | 497 (513)
  3 hours after administration | 938 (407)
  5 hours after administration: number analyzed (Participants) | 3
  5 hours after administration | 624 (235)
  8 hours after administration | 253 (103)

14. Primary Outcome: Non-Compartmental Pharmacokinetic (PK) Parameter of Tapentadol Area Under the Concentration-Time Curve (AUC 0-15) After a Single Dose of Tapentadol in Adolescent Participants (Age 12 to Less Than 18 Years).
Description: Serum samples for pharmacokinetic analysis were obtained using frequent sampling techniques in participants 12 years to less than 18 years of age.
  Serum samples (frequent sampling) were drawn at 0.25, 0.5, 1, 2, 4, 6, 11, and 15 hours.
  The Area Under the Curve (AUC) from dose to 15 hours (AUC 0-15) is a summary measure of data from each pharmacokinetic blood sample taken over the 15 hour time period.
  The area is that below the line fitted to the data points.
Time Frame: up to 15 hours
Population: The protocol planned that this analysis would only be performed for the adolescent participants.
Measure: Mean (Full Range); unit: ng*hr/mL
Groups:
- Tapentadol Non-Compartmental PK Parameter: AUC: Single Dose of Tapentadol Oral Solution in Adolescents Age 12 to Less Than 18 Years. Tapentadol oral solution single dose (1mg/kg body weight).
Arm/Group | Tapentadol Non-Compartmental PK Parameter: AUC
Number analyzed (Participants) | 18
ng*hr/mL | 302 [218 to 636]

15. Secondary Outcome: Respiratory Rate Assessments
Description: Respiratory rate assessments were performed at pre-defined times during the 15 hour period following investigational medicinal product intake.
  Pre-surgery data for these participants is also given from the enrollment Visit (Visit 1).
Time Frame: Enrollment Visit; 15 hours post-dose
Population: The protocol pre-specified that the young and very young children will be reported as one group.
  (Adolescents Group at and after 2 hours: N=20; Older Children Group at 30 minutes and 1 hour N=27, at 2 hours N=24, and at and after 4 hours N=22; Young and Very Young Children Group at and after 4 hours: N=16).
Measure: Mean (Standard Deviation); unit: breaths per minute
Groups:
- Respiratory Rates: Adolescents: Single Dose of Tapentadol Oral Solution in Adolescents Age 12 to Less Than 18 Years. Tapentadol oral solution single dose (1mg/kg body weight).
- Respiratory Rates: Older Children: Single Dose of Tapentadol Oral Solution in Children Age 6 to Less Than 12 Years. Tapentadol oral solution single dose (1mg/kg body weight).
- Respiratory Rates: Young and Very Young Children: Single Dose of Tapentadol Oral Solution in Children Age 2 to Less Than 6 Years. Tapentadol oral solution single dose (1mg/kg body weight).
Arm/Group | Respiratory Rates: Adolescents | Respiratory Rates: Older Children | Respiratory Rates: Young and Very Young Children
Number analyzed (Participants) | 21 | 28 | 17
breaths per minute
  Visit 1 | 17.8 (3.2) | 18.4 (3.1) | 25.1 (3.4)
  Pre-dose | 16.4 (2.5) | 19.2 (2.5) | 25.1 (3.3)
  15 minutes post-dose | 16.8 (2.6) | 19.7 (2.5) | 24.0 (3.1)
  30 minutes post-dose | 17.5 (2.5) | 19.4 (2.4) | 22.6 (4.3)
  1 hours post-dose | 15.9 (2.3) | 19.0 (2.0) | 21.8 (3.5)
  2 hours post-dose | 17.3 (2.8) | 19.3 (2.5) | 22.5 (3.3)
  4 hours post-dose | 16.4 (2.1) | 19.5 (2.8) | 22.5 (2.1)
  6 hours post-dose | 16.9 (2.9) | 19.0 (3.8) | 22.1 (3.5)
  11 hours post-dose | 17.4 (3.6) | 18.4 (2.9) | 22.4 (3.4)
  15 hours post-dose | 16.1 (2.5) | 17.3 (3.0) | 21.1 (3.9)

16. Secondary Outcome: Oxygen Saturation Assessments
Description: Oxygen saturation assessments were performed at pre-defined times during the 15 hour period following investigational medicinal product intake.
  Oxygen saturation was assessed using pulse oximetry. The uppermost value is 100%.
  Pre-surgery data for these participants is also given from the enrollment Visit (Visit 1).
Time Frame: Enrollment Visit; 15 hours post-dose
Population: The protocol pre-specified that the young and very young children will be reported as one group.
  (Adolescents Group at and after 2 hours: N=20; Older Children Group at 30 minutes and 1 hour N=27, at 2 hours N=24, at and after 4 hours N=22; Young and Very Young Children Group at and after 4 hours: N=16).
Measure: Mean (Standard Deviation); unit: percentage of oxygen saturation
Groups:
- Oxygen Saturation: Adolescents: Single Dose of Tapentadol Oral Solution in Adolescents Age 12 to Less Than 18 Years. Tapentadol oral solution single dose (1mg/kg body weight).
- Oxygen Saturation: Older Children: Single Dose of Tapentadol Oral Solution in Children Age 6 to Less Than 12 Years. Tapentadol oral solution single dose (1mg/kg body weight).
- Oxygen Saturation: Young and Very Young Children: Single Dose of Tapentadol Oral Solution in Children Age 2 to Less Than 6 Years. Tapentadol oral solution single dose (1mg/kg body weight).
Arm/Group | Oxygen Saturation: Adolescents | Oxygen Saturation: Older Children | Oxygen Saturation: Young and Very Young Children
Number analyzed (Participants) | 21 | 28 | 17
percentage of oxygen saturation
  Visit 1 | 97.8 (1.1) | 97.4 (1.7) | 97.4 (1.4)
  Pre-dose | 97.7 (1.4) | 96.7 (1.4) | 96.8 (1.0)
  15 minutes post-dose | 97.3 (1.2) | 96.8 (1.3) | 96.5 (1.9)
  30 minutes post-dose | 97.0 (1.4) | 96.4 (1.3) | 96.8 (1.6)
  1 hour post-dose | 97.3 (1.2) | 96.0 (1.6) | 96.2 (2.0)
  2 hours post-dose | 97.1 (1.3) | 95.8 (1.4) | 95.8 (1.7)
  4 hours post-dose | 96.9 (1.4) | 96.5 (1.2) | 96.5 (1.5)
  6 hours post-dose | 97.1 (1.5) | 96.7 (1.3) | 96.7 (1.7)
  11 hours post-dose | 96.8 (1.4) | 96.8 (1.4) | 96.4 (1.5)
  15 hours post-dose | 96.7 (1.0) | 96.5 (1.4) | 97.1 (1.5)

17. Secondary Outcome: Systolic and Diastolic Blood Pressure Assessments
Description: Systolic and Diastolic blood pressure assessments were performed at pre-defined times during the 15 hour period following investigational medicinal product intake.
  Pre-surgery data for these participants is also given from the enrollment Visit (Visit 1).
Time Frame: Enrollment Visit; 15 hours post-dose
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Blood Pressure: Adolescents: Single Dose of Tapentadol Oral Solution in Adolescents Age 12 to Less Than 18 Years. Tapentadol oral solution single dose (1mg/kg body weight).
- Blood Pressure: Older Children: Single Dose of Tapentadol Oral Solution in Children Age 6 to Less Than 12 Years. Tapentadol oral solution single dose (1mg/kg body weight).
- Blood Pressure: Young and Very Young Children: Single Dose of Tapentadol Oral Solution in Children Age 2 to Less Than 6 Years. Tapentadol oral solution single dose (1mg/kg body weight).
Arm/Group | Blood Pressure: Adolescents | Blood Pressure: Older Children | Blood Pressure: Young and Very Young Children
Number analyzed (Participants) | 21 | 28 | 17
mmHg
  Visit 1 Enrollment Systolic blood pressure | 110.2 (9.0) | 103.8 (9.6) | 98.7 (7.0)
  Pre-dose Systolic Blood Pressure | 122.9 (13.9) | 107.1 (9.1) | 105.1 (15.6)
  15 minutes post-dose Systolic Blood Pressure | 126.9 (17.7) | 104.1 (8.3) | 101.8 (7.5)
  30 minutes post-dose Systolic Blood Pressure | 126.8 (17.9) | 104.1 (7.2) | 100.1 (6.2)
  1 hour post-dose Systolic Blood Pressure | 127.0 (17.7) | 104.0 (9.6) | 97.6 (7.6)
  2 hours post-dose Systolic Blood Pressure | 124.9 (16.7) | 103.9 (8.2) | 98.4 (6.6)
  4 hours post-dose Systolic Blood Pressure | 122.8 (13.9) | 104.8 (10.5) | 100.1 (7.4)
  6 hours post-dose Systolic Blood Pressure | 116.8 (14.1) | 106.7 (7.9) | 102.0 (8.5)
  11 hours post-dose Systolic Blood Pressure | 115.1 (11.2) | 102.0 (9.1) | 99.4 (14.2)
  15 hours post-dose Systolic Blood Pressure | 113.8 (14.2) | 100.3 (8.7) | 93.3 (9.9)
  Visit 1 Enrollment Diastolic blood pressure | 66.5 (9.0) | 66.3 (8.3) | 62.8 (5.3)
  Pre-dose Diastolic blood pressure | 74.8 (11.8) | 64.2 (9.4) | 65.6 (11.2)
  15 minutes post-dose Diastolic blood pressure | 78.9 (15.7) | 62.4 (7.8) | 62.4 (7.7)
  30 minutes post-dose Diastolic blood pressure | 76.1 (12.0) | 61.3 (5.7) | 60.2 (6.1)
  1 hour post-dose Diastolic blood pressure | 77.6 (13.0) | 61.1 (7.1) | 59.6 (6.9)
  2 hours post-dose Diastolic blood pressure | 74.7 (13.4) | 59.7 (7.0) | 59.7 (7.4)
  4 hours post-dose Diastolic blood pressure | 73.2 (12.1) | 60.0 (7.1) | 58.7 (5.9)
  6 hours post-dose Diastolic blood pressure | 66.0 (10.3) | 59.0 (8.3) | 58.8 (7.3)
  11 hours post-dose Diastolic blood pressure | 65.4 (8.4) | 54.6 (8.5) | 57.3 (11.2)
  15 hours post-dose Diastolic blood pressure | 67.1 (10.8) | 56.8 (8.5) | 57.0 (8.7)

18. Secondary Outcome: Change From Enrollment in 12-lead Electrocardiogram Parameters
Description: 12-lead electrocardiograms (ECG) were part of the planned safety assessments. 12-lead Electrocardiograms were performed prior at the enrollment visit after informed consent and at the discharge visit. The discharge visit was as per standard of care.
  The changes in ECG parameters are reported. Negative mean values indicate that the millisecond intervals decreased from the enrollment to the discharge visit. Positive mean values indicate that the millisecond intervals increased from the enrollment to the discharge visit. The Letters P,Q,R,S and T refer to specific medically defined points on an ECG tracing and correspond to specific heart activities.
Time Frame: Enrollment (pre-surgery); Discharge Visit
Population: The protocol pre-specified that the young and very young children will be reported as one group.
  (For older children N=27 at Visit 1)
Measure: Mean (Standard Deviation); unit: milliseconds
Groups:
- ECG Changes: Adolescents: Single Dose of Tapentadol Oral Solution in Children and Adolescents Age 12 to Less Than 18 Years. Tapentadol oral solution single dose (1mg/kg body weight).
- ECG Changes: Older Children: Single Dose of Tapentadol Oral Solution in Children and Adolescents Age 6 to Less Than 12 Years. Tapentadol oral solution single dose (1mg/kg body weight).
- ECG Changes: Young and Very Young Children: Single Dose of Tapentadol Oral Solution in Children and Adolescents Age 2 to Less Than 6 Years. Tapentadol oral solution single dose (1mg/kg body weight).
Arm/Group | ECG Changes: Adolescents | ECG Changes: Older Children | ECG Changes: Young and Very Young Children
Number analyzed (Participants) | 21 | 27 | 17
milliseconds
  QTcF change | -3.6 (16.4) | 15.7 (21.7) | 5.6 (20.7)
  QT Duration change | -8.0 (33.1) | 8.5 (32.0) | -4.1 (29.6)
  QRS Duration change | 0.5 (4.5) | -0.2 (4.7) | 0.5 (5.8)
  PR Duration change | -3.5 (11.7) | -1.8 (11.3) | -2.4 (12.6)
  RR Duration change | -32.2 (193.8) | -35.2 (156.5) | -48.1 (102.8)

19. Secondary Outcome: Change From Enrollment in 12-lead Electrocardiogram Heart Rate Parameter
Description: 12-lead Electrocardiograms (ECG) were part of the planned safety assessments. 12-lead Electrocardiograms were performed prior at the enrollment visit after informed consent and at the discharge visit. The discharge visit was as per standard of care.
  The changes in heart rate (beats per minute) parameters are reported per treatment group between the visits.
  A positive value indicates that the heart rate was higher at discharge than at enrollment.
Time Frame: Enrollment; Discharge Visit
Population: The protocol pre-specified that the young and very young children will be reported as one group.
  (For older children: N=27 at Visit 1)
Measure: Mean (Standard Deviation); unit: beats per minute
Groups:
- ECG Heart Rate Change: Adolescents: Single Dose of Tapentadol Oral Solution in Children and Adolescents Age 12 to Less Than 18 Years. Tapentadol oral solution single dose (1mg/kg body weight).
- ECG Heart Rate Change: Older Children: Single Dose of Tapentadol Oral Solution in Children and Adolescents Age 6 to Less Than 12 Years. Tapentadol oral solution single dose (1mg/kg body weight).
- ECG Heart Rate Change: Young and Very Young Children: Single Dose of Tapentadol Oral Solution in Children and Adolescents Age 2 to Less Than 6 Years. Tapentadol oral solution single dose (1mg/kg body weight).
Arm/Group | ECG Heart Rate Change: Adolescents | ECG Heart Rate Change: Older Children | ECG Heart Rate Change: Young and Very Young Children
Number analyzed (Participants) | 21 | 28 | 17
beats per minute | 2.0 (16.4) | 4.3 (16.2) | 10.7 (16.4)

20. Primary Outcome: Non-Compartmental Pharmacokinetic (PK) Parameter: Cmax (Maximum Concentration) of Tapentadol After a Single Dose of Tapentadol in Adolescents (Age 12 to Less Than 18 Years).
Description: Serum samples for pharmacokinetic analysis were obtained using frequent sampling techniques in participants 12 years to less than 18 years of age.
  Serum samples (frequent sampling) were drawn at 0.25, 0.5, 1, 2, 4, 6, 11, and 15 hours. The concentration of tapentadol (active drug) is assessed during absorption and distribution.
  The maximum concentration is derived from the Area Under the Curve, from dose to 15 hours (AUC 0-15). It is the highest amount of active drug observed in the blood sample
Time Frame: up to 15 hours
Population: The protocol planned that this analysis would only be performed for the adolescent participants.
Measure: Mean (Standard Error); unit: nanograms/millilitre
Groups:
- Tapentadol Non-Compartmental PK Parameter: Cmax: Single Dose of Tapentadol Oral Solution in Adolescents Age 12 to Less Than 18 Years. Tapentadol oral solution single dose (1mg/kg body weight).
Arm/Group | Tapentadol Non-Compartmental PK Parameter: Cmax
Number analyzed (Participants) | 18
nanograms/millilitre | 67.5 (26.3)

21. Secondary Outcome: Treatment Emergent Adverse Events by Intensity
Description: The intensity of all treatment emergent adverse events (TEAEs) were scored by the investigator. Treatment emergent adverse events were those adverse events documented from the time of investigational medicinal product (IMP), study drug, up to 48 hours post dosing.
  The clinical "intensity" of an adverse event was classified as:
  * Mild: Signs and symptoms that can be easily tolerated. Symptoms can be ignored and disappear when the subject is distracted.
  * Moderate: Symptoms cause discomfort but are tolerable; they cannot be ignored and affect concentration.
  * Severe: Symptoms which affect usual daily activity.
  For adverse events where the intensity changes over time, the maximum intensity observed was documented.
Time Frame: Baseline; 48 hours post dosing
Population: The protocol pre-specified that the young and very young children will be reported as one group.
Measure: Number; unit: number of events
Groups:
- Number of TEAEs: Adolescents: Tapentadol oral solution single dose (1mg/kg body weight). Participants aged 12 years and less than 18 years of age.
- Number of TEAEs: Older Children: Tapentadol oral solution single dose (1mg/kg body weight). Participants aged 6 years and less than 12 years of age.
- Number of TEAEs: Young and Very Young Children: Tapentadol oral solution single dose (1mg/kg body weight). Participants aged 2 years and less than 6 years of age.
Arm/Group | Number of TEAEs: Adolescents | Number of TEAEs: Older Children | Number of TEAEs: Young and Very Young Children
Number analyzed (Participants) | 21 | 28 | 17
number of events
  Total number of TEAEs | 22 | 33 | 11
  Total number of mild TEAEs | 10 | 16 | 10
  Total number of moderate TEAEs | 12 | 17 | 1

22. Secondary Outcome: Intake of Additional Analgesic Medication During the Trial
Description: Number of participants with intakes of supplemental analgesic medication between investigational medicinal product (IMP) intake and Site Discharge grouped according to preparation taken (non-opioid/opioid).
Time Frame: Baseline; 15 hours post dosing
Population: The protocol pre-specified that the young and very young children will be reported as one group.
Measure: Number; unit: participants
Groups:
- Adolescents With Supplementary Analgesic: Single Dose of Tapentadol Oral Solution in Adolescents Age 12 to Less Than 18 Years. Tapentadol oral solution single dose (1mg/kg body weight).
- Older Children With Supplementary Analgesic: Single Dose of Tapentadol Oral Solution in Children Age 6 to Less Than 12 Years. Tapentadol oral solution single dose (1mg/kg body weight).
- Young and Very Young Children With Supplementary Analgesic: Single Dose of Tapentadol Oral Solution in Children Age 2 to Less Than 6 Years. Tapentadol oral solution single dose (1mg/kg body weight).
Arm/Group | Adolescents With Supplementary Analgesic | Older Children With Supplementary Analgesic | Young and Very Young Children With Supplementary Analgesic
Number analyzed (Participants) | 21 | 28 | 17
participants
  Supplemental analgesic medication taken | 12 | 18 | 15
  Supplemental opioid analgesic taken | 3 | 3 | 8
  Supplemental non-opioid analgesic taken | 12 | 18 | 15

23. Primary Outcome: Non-Compartmental Pharmacokinetic (PK) Parameter: Time to Maximum Concentration (Tmax) of Tapentadol After a Single Dose of Tapentadol in Adolescents (Age 12 to Less Than 18 Years).
Description: Serum samples for pharmacokinetic analysis were obtained using frequent sampling techniques in participants 12 years to less than 18 years of age.
  The time to maximum concentration is derived from the area under the curve from dose to 15 hours (AUC 0-15). The Tmax is the time after dosing at which the maximum concentration of the tapentadol (active drug) occurs.
  Serum samples (frequent sampling) were drawn at 0.25, 0.5, 1, 2, 4, 6, 11, and 15 hours.
Time Frame: up to 15 hours
Population: The protocol planned that this analysis would only be performed for the adolescent participants.
Measure: Mean (Standard Deviation); unit: hours
Groups:
- Tapentadol Non-Compartmental PK Parameter: Tmax: Tapentadol oral solution single dose (1mg/kg body weight) of participants aged 12 years to less than 18 years old.
Arm/Group | Tapentadol Non-Compartmental PK Parameter: Tmax
Number analyzed (Participants) | 18
hours | 1.4 (1.10)

24. Primary Outcome: Non-Compartmental Pharmacokinetic (PK) Parameter of Tapentadol-O-glucuronide Area Under the Concentration-Time Curve (AUC 0-15) After a Single Dose of Tapentadol in Adolescents (Age 12 to Less Than 18 Years).
Description: as for outcome 20
Time Frame: up to 15 hours
Population: The protocol planned that this analysis would only be performed for the adolescent participants.
Measure: Mean (Full Range); unit: ng*hr/mL
Groups:
- Tapentadol-O-glucuronide Non-Compartmental PK Parameter: AUC: Single Dose of Tapentadol Oral Solution in Adolescents Age 12 to Less Than 18 Years. Tapentadol oral solution single dose (1mg/kg body weight).
Arm/Group | Tapentadol-O-glucuronide Non-Compartmental PK Parameter: AUC
Number analyzed (Participants) | 18
ng*hr/mL | 7082 [4946 to 9689]

25. Primary Outcome: Non-Compartmental Pharmacokinetic (PK) Parameter: Cmax (Maximum Concentration) of Tapentadol-O-glucuronide After a Single Dose of Tapentadol in Adolescents (Age 12 to Less Than 18 Years).
Description: Tapentadol-O-glucuronide is the metabolite of tapentadol. Metabolites are sometimes referred to as "breakdown products". The body alters the administered medication to a metabolite so that it can be more easily or quickly removed from the body. Serum samples (frequent sampling) were drawn at 0.25, 0.5, 1, 2, 4, 6, 11, and 15 hours. The concentration of tapentadol-O-glucuronide (metabolite) is assessed to study absorption and distribution.
  The maximum concentration is derived from the Area Under the Curve, from dose to 15 hours (AUC 0-15). It is the highest amount of metabolite observed in the blood sample.
Time Frame: up to 15 hours
Population: The protocol planned that this analysis would only be performed for the adolescent participants.
Measure: Mean (Standard Error); unit: nanogramsg/millilitre
Groups:
- Tapentadol-O-glucuronide Non-Compartmental PK Parameter: Cmax: Single Dose of Tapentadol Oral Solution in Adolescents Age 12 to Less Than 18 Years. Tapentadol oral solution single dose (1mg/kg body weight).
Arm/Group | Tapentadol-O-glucuronide Non-Compartmental PK Parameter: Cmax
Number analyzed (Participants) | 18
nanogramsg/millilitre | 1487 (495)

26. Primary Outcome: Non-Compartmental Pharmacokinetic (PK) Parameter: Time to Maximum Concentration (Tmax) of Tapentadol-O-glucuronide After a Single Dose of Tapentadol in Adolescents (Age 12 to Less Than 18).
Description: Tapentadol-O-glucuronide is the metabolite of tapentadol. Metabolites are sometimes referred to as "breakdown products". The body alters the administered medication to a metabolite so that it can be more easily or quickly removed from the body. Serum samples for pharmacokinetic analysis were obtained using frequent sampling techniques in participants 12 years to less than 18 years of age. The time to maximum concentration is derived from the area under the curve from dose to 15 hours (AUC 0-15). The Tmax is the time after dosing at which the maximum concentration of the tapentadol-O-glucuronide (metabolite) occurs. Serum samples (frequent sampling) were drawn at 0.25, 0.5, 1, 2, 4, 6, 11, and 15 hours.
Time Frame: up to 15 hours
Population: The protocol planned that this analysis would only be performed for the adolescent participants.
Measure: Mean (Standard Deviation); unit: hours
Groups:
- Tapentadol-O-glucuronide Non-Compartmental PK Parameter: Tmax: Single Dose of Tapentadol Oral Solution in Adolescents Age 12 to Less Than 18 Years. Tapentadol oral solution single dose (1mg/kg body weight).
Arm/Group | Tapentadol-O-glucuronide Non-Compartmental PK Parameter: Tmax
Number analyzed (Participants) | 18
hours | 1.70 (1.19)

27. Secondary Outcome: Hematology Safety Laboratory Assessments: Hemoglobin Concentration
Description: The hemoglobin test is a commonly ordered blood test and was done as part of a complete blood count (CBC). It is routinely done before and after surgery to check for anemia, the presence of chronic kidney disease or other chronic medical problems. In the study there were 3 planned safety blood draws for routine blood tests: at Visit 1 (during the enrollment period, including surgery), at Visit 2 (prior to study drug administration) and at Visit 3 (prior to discharge from the hospital). The discharge visit was as per standard of care.
Time Frame: Enrollment Visit; Visit 2 and Discharge Visit
Population: The protocol pre-specified that the young and very young children will be reported as one group.
  (Adolescents Group at Visit 3: N=20 one participant with missing data; Young and Very Young Children Group at Visits 2 and 3: N=16 one participant with missing data at each of these visits).
Measure: Mean (Standard Deviation); unit: g/L
Groups:
- Hemoglobin Concentration: Adolescents: Single Dose of Tapentadol Oral Solution in Adolescents Age 12 to Less Than 18 Years. Tapentadol oral solution single dose (1mg/kg body weight).
- Hemoglobin Concentration: Older Children: Single Dose of Tapentadol Oral Solution in Children Age 6 to Less Than 12 Years. Tapentadol oral solution single dose (1mg/kg body weight).
- Hemoglobin Concentration: Young and Very Young Children: Single Dose of Tapentadol Oral Solution in Children Age 2 to Less Than 6 Years. Tapentadol oral solution single dose (1mg/kg body weight).
Arm/Group | Hemoglobin Concentration: Adolescents | Hemoglobin Concentration: Older Children | Hemoglobin Concentration: Young and Very Young Children
Number analyzed (Participants) | 21 | 28 | 17
g/L
  Visit 1 | 151.10 (13.82) | 140.04 (6.66) | 127.47 (7.60)
  Visit 2 | 145.67 (21.44) | 128.64 (7.88) | 121.75 (7.91)
  Visit 3 | 139.00 (19.20) | 126.54 (9.10) | 117.00 (7.63)

28. Secondary Outcome: Hematology Safety Laboratory Assessments: Hematocrit
Description: Hematocrit is a blood test that measures the percentage of the volume of whole blood that is made up of red blood cells (RBC). This measurement depends on the number of red blood cells and the size of red blood cells. In the study there were 3 planned safety blood draws for routine blood tests: at Visit 1 (during the enrollment period, including surgery), at Visit 2 (prior to study drug administration) and at Visit 3 (prior to discharge from the hospital). The discharge visit was as per standard of care.
Time Frame: Enrollment Visit; Visit 2 and Discharge Visit
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: fraction of blood volume
Groups:
- Hematocrit: Adolescents: Single Dose of Tapentadol Oral Solution in Adolescents Age 12 to Less Than 18 Years. Tapentadol oral solution single dose (1mg/kg body weight).
- Hematocrit: Older Children: Single Dose of Tapentadol Oral Solution in Children Age 6 to Less Than 12 Years. Tapentadol oral solution single dose (1mg/kg body weight).
- Hematocrit: Young and Very Young Children: Single Dose of Tapentadol Oral Solution in Children Age 2 to Less Than 6 Years. Tapentadol oral solution single dose (1mg/kg body weight).
Arm/Group | Hematocrit: Adolescents | Hematocrit: Older Children | Hematocrit: Young and Very Young Children
Number analyzed (Participants) | 21 | 28 | 17
fraction of blood volume
  Visit 1 | 0.436 (0.037) | 0.400 (0.018) | 0.368 (0.018)
  Visit 2 | 0.421 (0.060) | 0.372 (0.024) | 0.363 (0.023)
  Visit 3 | 0.402 (0.054) | 0.364 (0.025) | 0.356 (0.022)

29. Secondary Outcome: Hematology Safety Laboratory Assessments: Erythrocyte Mean Corpuscular Volume (Mean Corpuscular Volume)
Description: Erythrocyte Mean Corpuscular volume is a measurement of the average size of Red Blood Cells (RBC). It is also referred to as Mean Corpuscular Volume. In the study there were 3 planned safety blood draws for routine blood tests: at Visit 1 (during the enrollment period, including surgery), at Visit 2 (prior to study drug administration) and at Visit 3 (prior to discharge from the hospital). The discharge visit was as per standard of care.
Time Frame: Enrollment Visit; Visit 2 and Discharge Visit
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: fL
Groups:
- Mean Corpuscular Volume: Adolescents: Single Dose of Tapentadol Oral Solution in Adolescents Age 12 to Less Than 18 Years. Tapentadol oral solution single dose (1mg/kg body weight).
- Mean Corpuscular Volume: Older Children: Single Dose of Tapentadol Oral Solution in Children Age 6 to Less Than 12 Years. Tapentadol oral solution single dose (1mg/kg body weight).
- Mean Corpuscular Volume: Young and Very Young Children: Single Dose of Tapentadol Oral Solution in Children Age 2 to Less Than 6 Years. Tapentadol oral solution single dose (1mg/kg body weight).
Arm/Group | Mean Corpuscular Volume: Adolescents | Mean Corpuscular Volume: Older Children | Mean Corpuscular Volume: Young and Very Young Children
Number analyzed (Participants) | 21 | 28 | 17
fL
  Visit 1 | 86.1 (2.9) | 82.3 (3.1) | 79.6 (3.6)
  Visit 2 | 86.5 (2.1) | 83.1 (3.5) | 81.8 (3.7)
  Visit 3 | 86.9 (3.5) | 83.1 (3.5) | 82.7 (3.6)

30. Secondary Outcome: Hematology Safety Laboratory Assessments: Platelet Count
Description: Platelets are cell fragments that are vital for normal blood clotting. In the study there were 3 planned safety blood draws for routine blood tests: at Visit 1 (during the enrollment period, including surgery), at Visit 2 (prior to study drug administration) and at Visit 3 (prior to discharge from the hospital). The discharge visit was as per standard of care.
Time Frame: Enrollment Visit; Visit 2 and Discharge Visit
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: GI/L
Groups:
- Platelet Count: Adolescents: Single Dose of Tapentadol Oral Solution in Adolescents Age 12 to Less Than 18 Years. Tapentadol oral solution single dose (1mg/kg body weight).
- Platelet Count: Older Children: Single Dose of Tapentadol Oral Solution in Children Age 6 to Less Than 12 Years. Tapentadol oral solution single dose (1mg/kg body weight).
- Platelet Count: Young and Very Young Children: Single Dose of Tapentadol Oral Solution in Children Age 2 to Less Than 6 Years. Tapentadol oral solution single dose (1mg/kg body weight).
Arm/Group | Platelet Count: Adolescents | Platelet Count: Older Children | Platelet Count: Young and Very Young Children
Number analyzed (Participants) | 21 | 28 | 17
GI/L
  Visit 1 | 297.0 (59.8) | 347.1 (86.2) | 357.4 (67.5)
  Visit 2 | 266.1 (73.0) | 303.4 (73.9) | 312.6 (111.2)
  Visit 3 | 263.9 (57.9) | 316.9 (71.3) | 307.3 (50.0)

31. Secondary Outcome: Hematology Safety Laboratory Assessments: Leukocyte Concentration
Description: Leukocytes are also called white blood cells (WBC). These were measured to assess immune function. In the study there were 3 planned safety blood draws for routine blood tests: at Visit 1 (during the enrollment period, including surgery), at Visit 2 (prior to study drug administration) and at Visit 3 (prior to discharge from the hospital). The discharge visit was as per standard of care.
Time Frame: Enrollment Visit; Visit 2 and Discharge Visit
Population: The protocol pre-specified that the young and very young children will be reported as one group.
  (Adolescents Group at Visit 3: N=20 one participant with missing data; Young and Very Young Children Group at Visits 2 and 3: N=16 one participant with missing data at each visit).
Measure: Mean (Standard Deviation); unit: GI/L
Groups:
- Leukocyte Concentration: Adolescents: Single Dose of Tapentadol Oral Solution in Adolescents Age 12 to Less Than 18 Years. Tapentadol oral solution single dose (1mg/kg body weight).
- Leukocyte Concentration: Older Children: Single Dose of Tapentadol Oral Solution in Children Age 6 to Less Than 12 Years. Tapentadol oral solution single dose (1mg/kg body weight).
- Leukocyte Concentration: Young and Very Young Children: Single Dose of Tapentadol Oral Solution in Children Age 2 to Less Than 6 Years. Tapentadol oral solution single dose (1mg/kg body weight).
Arm/Group | Leukocyte Concentration: Adolescents | Leukocyte Concentration: Older Children | Leukocyte Concentration: Young and Very Young Children
Number analyzed (Participants) | 21 | 28 | 17
GI/L
  Visit 1 | 6.631 (1.682) | 7.594 (3.984) | 6.555 (1.278)
  Visit 2 | 8.537 (2.514) | 12.509 (4.209) | 10.751 (3.272)
  Visit 3 | 10.052 (3.253) | 14.806 (4.031) | 13.160 (2.907)

32. Secondary Outcome: Biochemistry Safety Laboratory Parameters: Blood Glucose Concentration
Description: A blood glucose test measures the amount of a sugar called glucose in blood. In the study there were 3 planned safety blood draws for routine blood tests: at Visit 1 (during the enrollment period, including surgery), at Visit 2 (prior to study drug administration) and at Visit 3 (prior to discharge from the hospital). The discharge visit was as per standard of care.
Time Frame: Enrollment Visit; Visit 2 and Discharge Visit
Population: The protocol pre-specified that the young and very young children will be reported as one group.
  (Adolescents Group at Visit 3: N=20 one participant with missing data; Young and Very Young Children Group at Visit 3: N=16 one participant with missing data).
Measure: Mean (Standard Deviation); unit: mmol/L
Groups:
- Blood Glucose Concentration: Adolescents: Single Dose of Tapentadol Oral Solution in Adolescents Age 12 to Less Than 18 Years. Tapentadol oral solution single dose (1mg/kg body weight).
- Blood Glucose Concentration: Older Children: Single Dose of Tapentadol Oral Solution in Children Age 6 to Less Than 12 Years. Tapentadol oral solution single dose (1mg/kg body weight).
- Blood Glucose Concentration: Young and Very Young Children: Single Dose of Tapentadol Oral Solution in Children Age 2 to Less Than 6 Years. Tapentadol oral solution single dose (1mg/kg body weight).
Arm/Group | Blood Glucose Concentration: Adolescents | Blood Glucose Concentration: Older Children | Blood Glucose Concentration: Young and Very Young Children
Number analyzed (Participants) | 21 | 28 | 17
mmol/L
  Visit 1 | 4.77 (0.51) | 4.81 (0.52) | 5.01 (1.38)
  Visit 2 | 5.10 (0.68) | 6.39 (1.49) | 5.89 (1.17)
  Visit 3 | 5.51 (0.90) | 5.69 (1.21) | 4.90 (0.54)

33. Secondary Outcome: Biochemistry Safety Laboratory Parameters: Blood Sodium Concentration
Description: Sodium is required by the body for the body to function properly. In the study there were 3 planned safety blood draws for routine blood tests: at Visit 1 (during the enrollment period, including surgery), at Visit 2 (prior to study drug administration) and at Visit 3 (prior to discharge from the hospital). The discharge visit was as per standard of care.
Time Frame: Enrollment Visit; Visit 2 and Discharge Visit
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: mmol/L
Groups:
- Blood Sodium Concentration: Adolescents: Single Dose of Tapentadol Oral Solution in Adolescents Age 12 to Less Than 18 Years. Tapentadol oral solution single dose (1mg/kg body weight).
- Blood Sodium Concentration: Older Children: Single Dose of Tapentadol Oral Solution in Children Age 6 to Less Than 12 Years. Tapentadol oral solution single dose (1mg/kg body weight).
- Blood Sodium Concentration: Young and Very Young Children: Single Dose of Tapentadol Oral Solution in Children Age 2 to Less Than 6 Years. Tapentadol oral solution single dose (1mg/kg body weight).
Arm/Group | Blood Sodium Concentration: Adolescents | Blood Sodium Concentration: Older Children | Blood Sodium Concentration: Young and Very Young Children
Number analyzed (Participants) | 21 | 28 | 17
mmol/L
  Visit 1 | 140.9 (1.4) | 140.4 (2.1) | 139.3 (1.3)
  Visit 2 | 140.3 (1.5) | 138.4 (2.6) | 139.1 (1.2)
  Visit 3 | 138.1 (1.2) | 138.7 (1.8) | 138.8 (1.9)

34. Secondary Outcome: Biochemistry Safety Laboratory Parameters: Blood Potassium Concentration
Description: Potassium is a mineral that the body needs to work normally. In the study there were 3 planned safety blood draws for routine blood tests: at Visit 1 (during the enrollment period, including surgery), at Visit 2 (prior to study drug administration) and at Visit 3 (prior to discharge from the hospital). The discharge visit was as per standard of care.
Time Frame: Enrollment Visit; Visit 2 and Discharge Visit
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: mmol/L
Groups:
- Blood Potassium Concentration: Adolescents: Single Dose of Tapentadol Oral Solution in Adolescents Age 12 to Less Than 18 Years. Tapentadol oral solution single dose (1mg/kg body weight).
- Blood Potassium Concentration: Older Children: Single Dose of Tapentadol Oral Solution in Children Age 6 to Less Than 12 Years. Tapentadol oral solution single dose (1mg/kg body weight).
- Blood Potassium Concentration: Young and Very Young Children: Single Dose of Tapentadol Oral Solution in Children Age 2 to Less Than 6 Years. Tapentadol oral solution single dose (1mg/kg body weight).
Arm/Group | Blood Potassium Concentration: Adolescents | Blood Potassium Concentration: Older Children | Blood Potassium Concentration: Young and Very Young Children
Number analyzed (Participants) | 21 | 28 | 17
mmol/L
  Visit 1 | 4.20 (0.31) | 4.20 (0.32) | 4.09 (0.33)
  Visit 2 | 3.90 (0.36) | 3.83 (0.32) | 4.04 (0.36)
  Visit 3 | 3.94 (0.26) | 3.93 (0.29) | 3.93 (0.27)

35. Secondary Outcome: Biochemistry Safety Laboratory Parameters: Blood Calcium Concentration
Description: All cells need calcium in order to function. In the study there were 3 planned safety blood draws for routine blood tests. In the study there were 3 planned safety blood draws for routine blood tests: at Visit 1 (during the enrollment period, including surgery), at Visit 2 (prior to study drug administration) and at Visit 3 (prior to discharge from the hospital). The discharge visit was as per standard of care.
Time Frame: Enrollment Visit; Visit 2 and Discharge Visit
Population: The protocol pre-specified that the young and very young children will be reported as one group.
  (Adolescents Group at Visit 3: N=20 one participant with missing data; Older children Group at Visit 2: N=27 one participant with missing data; Young and Very Young Children Group at Visit 3: N=16 one participant with missing data).
Measure: Mean (Standard Deviation); unit: mmol/L
Groups:
- Blood Calcium Concentration: Adolescents: Single Dose of Tapentadol Oral Solution in Adolescents Age 12 to Less Than 18 Years. Tapentadol oral solution single dose (1mg/kg body weight).
- Blood Calcium Concentration: Older Children: Single Dose of Tapentadol Oral Solution in Children Age 6 to Less Than 12 Years. Tapentadol oral solution single dose (1mg/kg body weight).
- Blood Calcium Concentration: Young and Very Young Children: Single Dose of Tapentadol Oral Solution in Children Age 2 to Less Than 6 Years. Tapentadol oral solution single dose (1mg/kg body weight).
Arm/Group | Blood Calcium Concentration: Adolescents | Blood Calcium Concentration: Older Children | Blood Calcium Concentration: Young and Very Young Children
Number analyzed (Participants) | 21 | 28 | 17
mmol/L
  Visit 1 | 2.455 (0.065) | 2.482 (0.100) | 2.519 (0.055)
  Visit 2 | 2.268 (0.166) | 2.267 (0.108) | 2.343 (0.160)
  Visit 3 | 2.359 (0.104) | 2.266 (0.157) | 2.369 (0.123)

36. Secondary Outcome: Biochemistry Safety Laboratory Parameters: Blood Chloride Concentration
Description: Chloride with other electrolytes help keep the proper balance of body fluids and maintain the body's acid-base balance. In the study there were 3 planned safety blood draws for routine blood tests: at Visit 1 (during the enrollment period, including surgery), at Visit 2 (prior to study drug administration) and at Visit 3 (prior to discharge from the hospital). The discharge visit was as per standard of care
Time Frame: Enrollment Visit; Visit 2 and Discharge Visit
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: mmol/L
Groups:
- Blood Chloride Concentration: Adolescents: Single Dose of Tapentadol Oral Solution in Adolescents Age 12 to Less Than 18 Years. Tapentadol oral solution single dose (1mg/kg body weight).
- Blood Chloride Concentration: Older Children: Single Dose of Tapentadol Oral Solution in Children Age 6 to Less Than 12 Years. Tapentadol oral solution single dose (1mg/kg body weight).
- Blood Chloride Concentration: Young and Very Young Children: Single Dose of Tapentadol Oral Solution in Children Age 2 to Less Than 6 Years. Tapentadol oral solution single dose (1mg/kg body weight).
Arm/Group | Blood Chloride Concentration: Adolescents | Blood Chloride Concentration: Older Children | Blood Chloride Concentration: Young and Very Young Children
Number analyzed (Participants) | 21 | 28 | 17
mmol/L
  Visit 1 | 103.3 (1.9) | 103.4 (2.2) | 103.8 (1.7)
  Visit 2 | 106.6 (2.2) | 104.9 (2.8) | 106.2 (3.0)
  Visit 3 | 103.0 (2.2) | 105.1 (2.6) | 105.1 (2.4)

37. Secondary Outcome: Biochemistry Safety Laboratory Parameters: Blood Phosphate Concentration
Description: Phosphate is needed by the body. This test was done to see how much phosphate is in the blood. In the study there were 3 planned safety blood draws for routine blood tests: at Visit 1 (during the enrollment period, including surgery), at Visit 2 (prior to study drug administration) and at Visit 3 (prior to discharge from the hospital). The discharge visit was as per standard of care.
Time Frame: Enrollment Visit; Visit 2 and Discharge Visit
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: mmol/L
Groups:
- Blood Phosphate Concentration: Adolescents: Single Dose of Tapentadol Oral Solution in Adolescents Age 12 to Less Than 18 Years. Tapentadol oral solution single dose (1mg/kg body weight).
- Blood Phosphate Concentration: Older Children: Single Dose of Tapentadol Oral Solution in Children Age 6 to Less Than 12 Years. Tapentadol oral solution single dose (1mg/kg body weight).
- Blood Phosphate Concentration: Young and Very Young Children: Single Dose of Tapentadol Oral Solution in Children Age 2 to Less Than 6 Years. Tapentadol oral solution single dose (1mg/kg body weight).
Arm/Group | Blood Phosphate Concentration: Adolescents | Blood Phosphate Concentration: Older Children | Blood Phosphate Concentration: Young and Very Young Children
Number analyzed (Participants) | 21 | 28 | 17
mmol/L
  Visit 1 | 1.384 (0.185) | 1.560 (0.146) | 1.689 (0.165)
  Visit 2 | 1.234 (0.194) | 1.248 (0.241) | 1.412 (0.179)
  Visit 3 | 1.500 (0.199) | 1.535 (0.178) | 1.611 (0.181)

38. Secondary Outcome: Biochemistry Safety Laboratory Parameters: Blood Urea Nitrogen (BUN) Concentration
Description: This test is to measure the amount of urea nitrogen in the blood. It was used to test liver and kidney function. In the study there were 3 planned safety blood draws for routine blood tests: at Visit 1 (during the enrollment period, including surgery), at Visit 2 (prior to study drug administration) and at Visit 3 (prior to discharge from the hospital). The discharge visit was as per standard of care.
Time Frame: Enrollment Visit; Visit 2 and Discharge Visit
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: mmol/L
Groups:
- BUN Concentration: Adolescents: Single Dose of Tapentadol Oral Solution in Adolescents Age 12 to Less Than 18 Years. Tapentadol oral solution single dose (1mg/kg body weight).
- BUN Concentration: Older Children: Single Dose of Tapentadol Oral Solution in Children Age 6 to Less Than 12 Years. Tapentadol oral solution single dose (1mg/kg body weight).
- BUN Concentration: Young and Very Young Children: Single Dose of Tapentadol Oral Solution in Children Age 2 to Less Than 6 Years. Tapentadol oral solution single dose (1mg/kg body weight).
Arm/Group | BUN Concentration: Adolescents | BUN Concentration: Older Children | BUN Concentration: Young and Very Young Children
Number analyzed (Participants) | 21 | 28 | 17
mmol/L
  Visit 1 | 4.55 (1.19) | 4.47 (1.30) | 5.15 (1.19)
  Visit 2 | 4.54 (1.32) | 4.38 (0.95) | 4.19 (0.93)
  Visit 3 | 3.88 (0.98) | 4.31 (1.21) | 4.11 (0.82)

39. Secondary Outcome: Biochemistry Safety Laboratory Parameters: Creatinine Concentration
Description: Creatinine is removed from the body entirely by the kidneys. If kidney function is not normal, creatinine level increases in the blood. In the study there were 3 planned safety blood draws for routine blood tests. In the study there were 3 planned safety blood draws for routine blood tests: at Visit 1 (during the enrollment period, including surgery), at Visit 2 (prior to study drug administration) and at Visit 3 (prior to discharge from the hospital). The discharge visit was as per standard of care.
Time Frame: Enrollment Visit; Visit 2 and Discharge Visit
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: µmol/L
Groups:
- Creatinine Concentration: Adolescents: Single Dose of Tapentadol Oral Solution in Adolescents Age 12 to Less Than 18 Years. Tapentadol oral solution single dose (1mg/kg body weight).
- Creatinine Concentration: Older Children: Single Dose of Tapentadol Oral Solution in Children Age 6 to Less Than 12 Years. Tapentadol oral solution single dose (1mg/kg body weight).
- Creatinine Concentration: Young and Very Young Children: Single Dose of Tapentadol Oral Solution in Children Age 2 to Less Than 6 Years. Tapentadol oral solution single dose (1mg/kg body weight).
Arm/Group | Creatinine Concentration: Adolescents | Creatinine Concentration: Older Children | Creatinine Concentration: Young and Very Young Children
Number analyzed (Participants) | 21 | 28 | 17
µmol/L
  Visit 1 | 73.3 (14.7) | 49.5 (6.2) | 35.6 (4.8)
  Visit 2 | 67.8 (15.1) | 44.1 (9.3) | 31.6 (6.7)
  Visit 3 | 68.6 (16.2) | 41.5 (8.0) | 33.0 (5.8)

40. Secondary Outcome: Biochemistry Safety Laboratory Parameters: Aspartate Aminotransferase (AST) Enzyme Activity
Description: AST is considered to be one of the two most important tests to detect liver injury. During liver damage the enzyme is released into the blood. In the study there were 3 planned safety blood draws for routine blood tests: at Visit 1 (during the enrollment period, including surgery), at Visit 2 (prior to study drug administration) and at Visit 3 (prior to discharge from the hospital). The discharge visit was as per standard of care.
Time Frame: Enrollment Visit; Visit 2 and Discharge Visit
Population: The protocol pre-specified that the young and very young children will be reported as one group.
  (Adolescents Group at Visit 3: N=20 one participant with missing data; Older children at Visits 2 and 3: N=26 two participants with missing data; Young and Very Young Children Group at Visits 1 and 3: N=16 one participant with missing data).
Measure: Mean (Standard Deviation); unit: U/L
Groups:
- AST Activity: Adolescents: Single Dose of Tapentadol Oral Solution in Adolescents Age 12 to Less Than 18 Years. Tapentadol oral solution single dose (1mg/kg body weight).
- AST Activity: Older Children: Single Dose of Tapentadol Oral Solution in Children Age 6 to Less Than 12 Years. Tapentadol oral solution single dose (1mg/kg body weight).
- AST Activity: Young and Very Young Children: Single Dose of Tapentadol Oral Solution in Children Age 2 to Less Than 6 Years. Tapentadol oral solution single dose (1mg/kg body weight).
Arm/Group | AST Activity: Adolescents | AST Activity: Older Children | AST Activity: Young and Very Young Children
Number analyzed (Participants) | 21 | 28 | 17
U/L
  Visit 1 | 21.5 (5.1) | 27.9 (6.5) | 33.4 (3.8)
  Visit 2 | 21.6 (4.5) | 29.9 (5.1) | 37.9 (7.5)
  Visit 3 | 21.6 (12.9) | 30.2 (7.2) | 33.8 (4.4)

41. Secondary Outcome: Biochemistry Safety Laboratory Parameters: Triglycerides Concentration
Description: Triglycerides are a group of fat. Triglycerides were measured as part of metabolic and cardiac assessments. In the study there were 3 planned safety blood draws for routine blood tests: at Visit 1 (during the enrollment period, including surgery), at Visit 2 (prior to study drug administration) and at Visit 3 (prior to discharge from the hospital). The discharge visit was as per standard of care.
Time Frame: Enrollment Visit; Visit 2 and Discharge Visit
Population: The protocol pre-specified that the young and very young children will be reported as one group.
  (Adolescents Group at Visit 3: N=20 one participant data missing; Older children Visits 2 and 3: N=27 and N=26 one and two participant data missing; Young and Very Young Children Group at Visits 2 and 3: N=16 one participant data missing).
Measure: Mean (Standard Deviation); unit: mmol/L
Groups:
- Triglycerides Concentration: Adolescents: Single Dose of Tapentadol Oral Solution in Adolescents Age 12 to Less Than 18 Years. Tapentadol oral solution single dose (1mg/kg body weight).
- Triglycerides Concentration: Older Children: Single Dose of Tapentadol Oral Solution in Children Age 6 to Less Than 12 Years. Tapentadol oral solution single dose (1mg/kg body weight).
- Triglycerides Concentration: Young and Very Young Children: Single Dose of Tapentadol Oral Solution in Children Age 2 to Less Than 6 Years. Tapentadol oral solution single dose (1mg/kg body weight).
Arm/Group | Triglycerides Concentration: Adolescents | Triglycerides Concentration: Older Children | Triglycerides Concentration: Young and Very Young Children
Number analyzed (Participants) | 21 | 28 | 17
mmol/L
  Visit 1 | 1.118 (0.459) | 1.129 (0.495) | 1.223 (0.511)
  Visit 2 | 0.666 (0.318) | 0.499 (0.245) | 0.556 (0.173)
  Visit 3 | 0.634 (0.224) | 0.646 (0.225) | 0.789 (0.227)

42. Secondary Outcome: Biochemistry Safety Laboratory Parameters: Serum Albumin Concentration
Description: Albumin is a protein made by the liver. Albumin prevents fluid leaking into the tissues. Albumin also transports many small molecules. Serum albumin was measured in the clear liquid portion of the blood called serum. In the study there were 3 planned safety blood draws for routine blood tests: at Visit 1 (during the enrollment period, including surgery), at Visit 2 (prior to study drug administration) and at Visit 3 (prior to discharge from the hospital). The discharge visit was as per standard of care.
Time Frame: Enrollment Visit; Visit 2 and Discharge Visit
Population: The protocol pre-specified that the young and very young children will be reported as one group.
  (Adolescents Group at Visit 3: N=20 one participant with missing data; Older children N=27 at Visit 1; Young and Very Young Children Group at Visit 3: N=16 one participant with missing data).
Measure: Mean (Standard Deviation); unit: g/L
Groups:
- Albumin Concentration: Adolescents: Single Dose of Tapentadol Oral Solution in Adolescents Age 12 to Less Than 18 Years. Tapentadol oral solution single dose (1mg/kg body weight).
- Albumin Concentration: Older Children: Single Dose of Tapentadol Oral Solution in Children Age 6 to Less Than 12 Years. Tapentadol oral solution single dose (1mg/kg body weight).
- Albumin Concentration: Young and Very Young Children: Single Dose of Tapentadol Oral Solution in Children Age 2 to Less Than 6 Years. Tapentadol oral solution single dose (1mg/kg body weight).
Arm/Group | Albumin Concentration: Adolescents | Albumin Concentration: Older Children | Albumin Concentration: Young and Very Young Children
Number analyzed (Participants) | 21 | 28 | 17
g/L
  Visit 1 | 43.4 (2.5) | 43.4 (3.0) | 42.6 (2.4)
  Visit 2 | 38.4 (3.1) | 37.1 (2.5) | 38.9 (3.4)
  Visit 3 | 38.4 (2.8) | 37.2 (3.5) | 37.5 (3.3)

43. Secondary Outcome: Biochemistry Safety Laboratory Parameters: Urate in the Blood
Description: Uric acid (urate is the salt) is a chemical created when the body breaks down substances called purines. Most urate dissolves in blood and travels to the kidneys. From there, it passes out in the urine. The test is used to determine kidney function. In the study there were 3 planned safety blood draws for routine blood tests: at Visit 1 (during the enrollment period, including surgery), at Visit 2 (prior to study drug administration) and at Visit 3 (prior to discharge from the hospital). The discharge visit was as per standard of care.
Time Frame: Enrollment Visit; Visit 2 and Discharge Visit
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: µmol/L
Groups:
- Urate: Adolescents: Single Dose of Tapentadol Oral Solution in Adolescents Age 12 to Less Than 18 Years. Tapentadol oral solution single dose (1mg/kg body weight).
- Urate: Older Children: Single Dose of Tapentadol Oral Solution in Children Age 6 to Less Than 12 Years. Tapentadol oral solution single dose (1mg/kg body weight).
- Urate: Young and Very Young Children: Single Dose of Tapentadol Oral Solution in Children Age 2 to Less Than 6 Years. Tapentadol oral solution single dose (1mg/kg body weight).
Arm/Group | Urate: Adolescents | Urate: Older Children | Urate: Young and Very Young Children
Number analyzed (Participants) | 21 | 28 | 17
µmol/L
  Visit 1 | 301.62 (69.35) | 228.32 (41.87) | 214.82 (39.67)
  Visit 2 | 305.57 (85.12) | 225.39 (44.74) | 205.65 (34.51)
  Visit 3 | 291.45 (69.06) | 213.68 (57.96) | 195.94 (48.68)

44. Secondary Outcome: Biochemistry Safety Laboratory Parameters: Calculated Glomerular Filtration Rate
Description: Glomerular filtration rate (GFR) was done to check how well the kidneys are working. It estimates how much blood passes through the glomeruli in the kidney each minute. In the study there were 3 planned safety blood draws for routine blood tests: at Visit 1 (during the enrollment period, including surgery), at Visit 2 (prior to study drug administration) and at Visit 3 (prior to discharge from the hospital). The discharge visit was as per standard of care.
Time Frame: Enrollment Visit; Visit 2 and Discharge Visit
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Groups:
- Glomerular Filtration Rate: Adolescents: Single Dose of Tapentadol Oral Solution in Adolescents Age 12 to Less Than 18 Years. Tapentadol oral solution single dose (1mg/kg body weight).
- Glomerular Filtration Rate: Older Children: Single Dose of Tapentadol Oral Solution in Children Age 6 to Less Than 12 Years. Tapentadol oral solution single dose (1mg/kg body weight).
- Glomerular Filtration Rate: Young and Very Young Children: Single Dose of Tapentadol Oral Solution in Children Age 2 to Less Than 6 Years. Tapentadol oral solution single dose (1mg/kg body weight).
Arm/Group | Glomerular Filtration Rate: Adolescents | Glomerular Filtration Rate: Older Children | Glomerular Filtration Rate: Young and Very Young Children
Number analyzed (Participants) | 21 | 28 | 17
mL/min/1.73m^2
  Visit 1 | 133.6 (20.7) | 133.9 (16.6) | 141.5 (18.4)
  Visit 2 | 146.6 (25.2) | 155.1 (38.0) | 166.9 (42.5)
  Visit 3 | 142.6 (23.3) | 158.7 (31.5) | 164.0 (37.3)

45. Secondary Outcome: Biochemistry Safety Laboratory Parameters: Urine Specific Gravity
Description: This test was used to test for the water balance and urine concentration. A urine sample was tested right away. A dipstick with a color-sensitive pad was used. The color the dipstick changes and the specific gravity of the urine was read off the color chart. In the study there were 2 planned safety urine collections. At Visit 1 in the enrollment period, after consent and assent obtained. The second sample was obtained at Visit 3 prior to discharge from the hospital. The discharge visit was as per standard of care.
Time Frame: Enrollment Visit and Discharge Visit
Population: The protocol pre-specified that the young and very young children will be reported as one group.
  (Young and Very Young Children Group at Visits 1: N=9 thus 8 participants with missing data; at Visit 3: N=7 thus 10 participants with missing data).
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Specific Gravity Urine: Adolescents: Single Dose of Tapentadol Oral Solution in Adolescents Age 12 to Less Than 18 Years. Tapentadol oral solution single dose (1mg/kg body weight).
- Specific Gravity Urine: Older Children: Single Dose of Tapentadol Oral Solution in Children Age 6 to Less Than 12 Years. Tapentadol oral solution single dose (1mg/kg body weight).
- Specific Gravity Urine: Young and Very Young Children: Single Dose of Tapentadol Oral Solution in Children Age 2 to Less Than 6 Years. Tapentadol oral solution single dose (1mg/kg body weight).
Arm/Group | Specific Gravity Urine: Adolescents | Specific Gravity Urine: Older Children | Specific Gravity Urine: Young and Very Young Children
Number analyzed (Participants) | 21 | 28 | 17
units on a scale
  Visit 1 | 1.025 (0.007) | 1.024 (0.004) | 1.021 (0.007)
  Visit 3 | 1.022 (0.007) | 1.024 (0.004) | 1.024 (0.002)

46. Secondary Outcome: Biochemistry Safety Laboratory Parameters: Urine pH (Acid, Alkalinity) Test
Description: A urine sample was tested right away. A dipstick made with a color-sensitive pad was used. The color indicated the acidity of the urine. In the study there were 2 planned safety urine collections. At Visit 1 in the enrollment period, after consent and assent obtained. The second sample was obtained at Visit 3 prior to discharge from the hospital. The discharge visit was as per standard of care.
Time Frame: Enrollment Visit and Discharge Visit
Population: as for outcome 45
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Urine pH: Adolescents: Single Dose of Tapentadol Oral Solution in Adolescents Age 12 to Less Than 18 Years. Tapentadol oral solution single dose (1mg/kg body weight).
- Urine pH: Older Children: Single Dose of Tapentadol Oral Solution in Children Age 6 to Less Than 12 Years. Tapentadol oral solution single dose (1mg/kg body weight).
- Urine pH: Young and Very Young Children: Single Dose of Tapentadol Oral Solution in Children Age 2 to Less Than 6 Years. Tapentadol oral solution single dose (1mg/kg body weight).
Arm/Group | Urine pH: Adolescents | Urine pH: Older Children | Urine pH: Young and Very Young Children
Number analyzed (Participants) | 21 | 28 | 17
units on a scale
  Visit 1 | 6.2 (0.5) | 6.5 (0.4) | 6.2 (0.6)
  Visit 3 | 6.1 (0.2) | 6.2 (0.4) | 6.4 (0.9)

47. Secondary Outcome: Biochemistry Safety Laboratory Parameters: Liver Function Test - Alanine Aminotransferase (ALT) Enzyme Activity
Description: This test was done in combination with other tests (such as AST, ALP, and bilirubin) to diagnose and monitor the liver function. In the study there were 3 planned safety blood draws for routine blood tests. In the study there were 3 planned safety blood draws for routine blood tests: at Visit 1 (during the enrollment period, including surgery), at Visit 2 (prior to study drug administration) and at Visit 3 (prior to discharge from the hospital). The discharge visit was as per standard of care.
Time Frame: Enrollment Visit, Visit 2 and Discharge Visit
Population: The protocol pre-specified that the young and very young children will be reported as one group.
  (Adolescents Group at Visit 3: N=19 two participants with missing data; Young and Very Young Children Group at Visit 3: N=16 one participant with missing data).
Measure: Mean (Standard Deviation); unit: U/L
Groups:
- ALT Activity: Adolescents: Single Dose of Tapentadol Oral Solution in Adolescents Age 12 to Less Than 18 Years. Tapentadol oral solution single dose (1mg/kg body weight).
- ALT Activity: Older Children: Single Dose of Tapentadol Oral Solution in Children Age 6 to Less Than 12 Years. Tapentadol oral solution single dose (1mg/kg body weight).
- ALT Activity: Young & Very Young Children: Single Dose of Tapentadol Oral Solution in Children Age 2 to Less Than 6 Years. Tapentadol oral solution single dose (1mg/kg body weight).
Arm/Group | ALT Activity: Adolescents | ALT Activity: Older Children | ALT Activity: Young & Very Young Children
Number analyzed (Participants) | 21 | 28 | 17
U/L
  Visit 1 | 16.2 (6.3) | 15.9 (4.1) | 16.4 (3.4)
  Visit 2 | 14.1 (4.6) | 15.7 (3.4) | 17.9 (5.3)
  Visit 3 | 14.2 (4.5) | 15.4 (3.4) | 17.1 (4.1)

48. Secondary Outcome: Biochemistry Safety Laboratory Parameters: Liver Function Test - Gamma-Glutamyl Transferase (GGT) Enzyme Activity
Description: The gamma-glutamyl transferase (GGT) test was used in combination with the alkaline phosphatase (ALP) test. Both ALP and GGT can be elevated in bile duct or liver complications. In the study there were 3 planned safety blood draws for routine blood tests: at Visit 1 (during the enrollment period, including surgery), at Visit 2 (prior to study drug administration) and at Visit 3 (prior to discharge from the hospital). The discharge visit was as per standard of care.
Time Frame: Enrollment Visit, Visit 2 and Discharge Visit
Population: The protocol pre-specified that the young and very young children will be reported as one group.
  (Adolescents Group at Visit 2 and 3: N=20 one participant with missing data; Older Children at Visit 2: N=27 one participant with missing data; Young and Very Young Children Group at Visit 2: N=16 one participant with missing data).
Measure: Mean (Standard Deviation); unit: U/L
Groups:
- GGT Activity: Adolescents: Single Dose of Tapentadol Oral Solution in Adolescents Age 12 to Less Than 18 Years. Tapentadol oral solution single dose (1mg/kg body weight).
- GGT Activity: Older Children: Single Dose of Tapentadol Oral Solution in Children Age 6 to Less Than 12 Years. Tapentadol oral solution single dose (1mg/kg body weight).
- GGT Activity: Young & Very Young Children: Single Dose of Tapentadol Oral Solution in Children Age 2 to Less Than 6 Years. Tapentadol oral solution single dose (1mg/kg body weight).
Arm/Group | GGT Activity: Adolescents | GGT Activity: Older Children | GGT Activity: Young & Very Young Children
Number analyzed (Participants) | 21 | 28 | 17
U/L
  Visit 1 | 12.0 (4.0) | 10.6 (2.9) | 9.4 (1.7)
  Visit 2 | 10.4 (3.9) | 8.7 (2.0) | 8.6 (1.9)
  Visit 3 | 10.8 (4.2) | 8.8 (1.9) | 8.3 (2.0)

49. Secondary Outcome: Biochemistry Safety Laboratory Parameters: Liver Function Test - Bilirubin Concentration
Description: Old red blood cells are replaced by new blood cells every day. Bilirubin is made by the body when the old blood cells are removed. The concentration of bilirubin in the blood measures liver function. In the study there were 3 planned safety blood draws for routine blood tests: at Visit 1 (during the enrollment period, including surgery), at Visit 2 (prior to study drug administration) and at Visit 3 (prior to discharge from the hospital). The discharge visit was as per standard of care.
Time Frame: Enrollment Visit, Visit 2 and Discharge Visit
Population: The protocol pre-specified that the young and very young children will be reported as one group.
  (Adolescents-Visit 2 & 3: N=20 - 1 participant with data missing; Older Children-Visit 1 & 2: N=26 thus 2 participants with data missing; Young and Very Young Children-Visits 1 & 3: N=12 (5 with data missing) & at Visit 2 N=9 (8 with data missing).
Measure: Mean (Standard Deviation); unit: µmol/L
Groups:
- Bilirubin Concentration: Adolescents: Single Dose of Tapentadol Oral Solution in Adolescents Age 12 to Less Than 18 Years. Tapentadol oral solution single dose (1mg/kg body weight).
- Bilirubin Concentration: Older Children: Single Dose of Tapentadol Oral Solution in Children Age 6 to Less Than 12 Years. Tapentadol oral solution single dose (1mg/kg body weight).
- Bilirubin Concentration: Young & Very Young Children: Single Dose of Tapentadol Oral Solution in Children Age 2 to Less Than 6 Years. Tapentadol oral solution single dose (1mg/kg body weight).
Arm/Group | Bilirubin Concentration: Adolescents | Bilirubin Concentration: Older Children | Bilirubin Concentration: Young & Very Young Children
Number analyzed (Participants) | 21 | 28 | 17
µmol/L
  Visit 1 | 12.0 (7.0) | 6.8 (3.5) | 4.8 (1.8)
  Visit 2 | 10.9 (7.8) | 6.3 (2.3) | 3.7 (1.0)
  Visit 3 | 17.8 (10.8) | 9.3 (4.5) | 5.8 (2.6)

50. Secondary Outcome: Biochemistry Safety Laboratory Parameters: Liver Function Test - Lactate Dehydrogenase (LDH) Enzyme Activity
Description: Lactate Dehydrogenase (LDH) was used to check for tissue damage. In the study there were 3 planned safety blood draws for routine blood tests: at Visit 1 (during the enrollment period, including surgery), at Visit 2 (prior to study drug administration) and at Visit 3 (prior to discharge from the hospital). The discharge visit was as per standard of care.
Time Frame: Enrollment Visit, Visit 2 and Discharge Visit
Population: The protocol pre-specified that the young and very young children will be reported as one group.
  (Adolescents Group at Visit 3: N=20 one participant with missing data; Older Children at Visits 1 and 3: N=26 and at Visit 2 N=24 participants; Young and Very Young Children Group at Visits 1 and 3: N=16 participant with missing data).
Measure: Mean (Standard Deviation); unit: U/L
Groups:
- LDH Activity: Adolescents: Single Dose of Tapentadol Oral Solution in Adolescents Age 12 to Less Than 18 Years. Tapentadol oral solution single dose (1mg/kg body weight).
- LDH Activity: Older Children: Single Dose of Tapentadol Oral Solution in Children Age 6 to Less Than 12 Years. Tapentadol oral solution single dose (1mg/kg body weight).
- LDH Activity: Young & Very Young Children: Single Dose of Tapentadol Oral Solution in Children Age 2 to Less Than 6 Years. Tapentadol oral solution single dose (1mg/kg body weight).
Arm/Group | LDH Activity: Adolescents | LDH Activity: Older Children | LDH Activity: Young & Very Young Children
Number analyzed (Participants) | 21 | 28 | 17
U/L
  Visit 1 | 157.7 (23.0) | 210.5 (31.7) | 243.8 (23.3)
  Visit 2 | 154.5 (27.9) | 199.1 (27.2) | 256.3 (36.8)
  Visit 3 | 143.9 (28.8) | 197.8 (28.5) | 238.6 (24.6)

51. Secondary Outcome: Biochemistry Safety Laboratory Parameters: Blood Protein Concentration
Description: The test was done to verify kidney and liver function. It is done in combination with the albumin test. In the study there were 3 planned safety blood draws for routine blood tests: at Visit 1 (during the enrollment period, including surgery), at Visit 2 (prior to study drug administration) and at Visit 3 (prior to discharge from the hospital). The discharge visit was as per standard of care.
Time Frame: Enrollment Visit, Visit 2 and Discharge Visit
Population: The protocol pre-specified that the young and very young children will be reported as one group.
  (Adolescents Group at Visit 3: N=20 one participant with missing data; Older Children at Visit 2: N=27 one participant with missing data; Young and Very Young Children Group at Visit 3: N=16 one participant with missing data).
Measure: Mean (Standard Deviation); unit: g/L
Groups:
- Protein Concentration: Adolescents: Single Dose of Tapentadol Oral Solution in Adolescents Age 12 to Less Than 18 Years. Tapentadol oral solution single dose (1mg/kg body weight).
- Protein Concentration: Older Children: Single Dose of Tapentadol Oral Solution in Children Age 6 to Less Than 12 Years. Tapentadol oral solution single dose (1mg/kg body weight).
- Protein Concentration: Young & Very Young Children: Single Dose of Tapentadol Oral Solution in Children Age 2 to Less Than 6 Years. Tapentadol oral solution single dose (1mg/kg body weight).
Arm/Group | Protein Concentration: Adolescents | Protein Concentration: Older Children | Protein Concentration: Young & Very Young Children
Number analyzed (Participants) | 21 | 28 | 17
g/L
  Visit 1 | 72.3 (3.5) | 73.3 (4.4) | 68.6 (4.7)
  Visit 2 | 64.2 (4.6) | 61.8 (4.4) | 62.1 (4.9)
  Visit 3 | 64.9 (4.4) | 62.1 (5.5) | 61.8 (4.6)

52. Secondary Outcome: Biochemistry Safety Laboratory Parameters: Creatine Kinase (CK) Enzyme Activity
Description: The creatine kinase (CK) test was used to detect inflammation of muscles. The test was done in combination with other tests. In the study there were 3 planned safety blood draws for routine blood tests: at Visit 1 (during the enrollment period, including surgery), at Visit 2 (prior to study drug administration) and at Visit 3 (prior to discharge from the hospital). The discharge visit was as per standard of care.
Time Frame: Enrollment Visit, Visit 2 and Discharge Visit
Population: The protocol pre-specified that the young and very young children will be reported as one group.
  (Adolescents Group at Visit 3: N=20 one participant with missing data; Older children at Visit 1: N=27 (1 participant missing); Young and Very Young Children Group at Visit 3: N=16 one participant with missing data at this visit).
Measure: Mean (Standard Deviation); unit: U/L
Groups:
- CK Activity: Adolescents: Single Dose of Tapentadol Oral Solution in Adolescents Age 12 to Less Than 18 Years. Tapentadol oral solution single dose (1mg/kg body weight).
- CK Activity: Older Children: Single Dose of Tapentadol Oral Solution in Children Age 6 to Less Than 12 Years. Tapentadol oral solution single dose (1mg/kg body weight).
- CK Activity: Young & Very Young Children: Single Dose of Tapentadol Oral Solution in Children Age 2 to Less Than 6 Years. Tapentadol oral solution single dose (1mg/kg body weight).
Arm/Group | CK Activity: Adolescents | CK Activity: Older Children | CK Activity: Young & Very Young Children
Number analyzed (Participants) | 21 | 28 | 17
U/L
  Visit 1 | 126.0 (66.0) | 109.8 (31.7) | 133.4 (35.2)
  Visit 2 | 186.8 (216.2) | 283.3 (158.5) | 275.8 (87.5)
  Visit 3 | 264.6 (564.4) | 288.1 (214.8) | 203.6 (84.5)

53. Secondary Outcome: Biochemistry Safety Laboratory Parameters: Alkaline Phosphatase (ALP) Enzyme Activity
Description: The Alkaline Phosphatase activity was used to detect bone or hepatobiliary disease. In the study there were 3 planned safety blood draws for routine blood tests: at Visit 1 (during the enrollment period, including surgery), at Visit 2 (prior to study drug administration) and at Visit 3 (prior to discharge from the hospital). The discharge visit was as per standard of care.
Time Frame: Enrollment Visit, Visit 2 and Discharge Visit
Population: The protocol pre-specified that the young and very young children will be reported as one group.
  (Adolescents Group at Visit 2 and 3: N=20 one participant with missing data; Young and Very Young Children Group at Visits 3: N=16 one participant with missing data at this visit).
Measure: Mean (Standard Deviation); unit: U/L
Groups:
- ALP Activity: Adolescents: Single Dose of Tapentadol Oral Solution in Adolescents Age 12 to Less Than 18 Years. Tapentadol oral solution single dose (1mg/kg body weight).
- ALP Activity: Older Children: Single Dose of Tapentadol Oral Solution in Children Age 6 to Less Than 12 Years. Tapentadol oral solution single dose (1mg/kg body weight).
- ALP Activity: Young & Very Young Children: Single Dose of Tapentadol Oral Solution in Children Age 2 to Less Than 6 Years. Tapentadol oral solution single dose (1mg/kg body weight).
Arm/Group | ALP Activity: Adolescents | ALP Activity: Older Children | ALP Activity: Young & Very Young Children
Number analyzed (Participants) | 21 | 28 | 17
U/L
  Visit 1 | 124.7 (62.7) | 240.0 (50.8) | 230.1 (26.7)
  Visit 2 | 114.7 (53.9) | 207.5 (42.2) | 210.2 (31.5)
  Visit 3 | 107.6 (54.3) | 204.1 (46.7) | 199.2 (26.2)

54. Secondary Outcome: Biochemistry Safety Laboratory Parameters: Triacylglycerol Lipase (TL) Enzyme Activity
Description: A triacylglycerol lipase test was done to check for pancreatic function. In the study there were 3 planned safety blood draws for routine blood tests. In the study there were 3 planned safety blood draws for routine blood tests: at Visit 1 (during the enrollment period, including surgery), at Visit 2 (prior to investigational medicinal product administration) and at Visit 3 (prior to discharge from the hospital). The discharge visit was as per standard of care.
Time Frame: Enrollment Visit, Visit 2 and Discharge Visit
Population: The protocol pre-specified that the young and very young children will be reported as one group.
  (Adolescents Group at Visit 3: N=20 one participant with missing data; Older Children N=27 at Visit 1 one participant with missing data; Young and Very Young Children Group at Visit 3: N=16 one participant with missing data at visit).
Measure: Mean (Standard Deviation); unit: U/L
Groups:
- TL Activity: Adolescents: Single Dose of Tapentadol Oral Solution in Adolescents Age 12 to Less Than 18 Years. Tapentadol oral solution single dose (1mg/kg body weight).
- TL Activity: Older Children: Single Dose of Tapentadol Oral Solution in Children Age 6 to Less Than 12 Years. Tapentadol oral solution single dose (1mg/kg body weight).
- TL Activity: Young & Very Young Children: Single Dose of Tapentadol Oral Solution in Children Age 2 to Less Than 6 Years. Tapentadol oral solution single dose (1mg/kg body weight).
Arm/Group | TL Activity: Adolescents | TL Activity: Older Children | TL Activity: Young & Very Young Children
Number analyzed (Participants) | 21 | 28 | 17
U/L
  Visit 1 | 29.5 (10.5) | 30.3 (9.4) | 26.3 (8.7)
  Visit 2 | 22.7 (8.3) | 22.6 (8.8) | 19.6 (6.3)
  Visit 3 | 24.8 (18.3) | 22.2 (9.2) | 19.3 (6.0)

ADVERSE EVENTS:
Time Frame: Any adverse event that started on the intake of tapentadol up to 48 hours thereafter.
Description: For tapentadol oral solution, the therapeutic reach is defined as 48 hours after intake.
  The age groups reported were prespecified in the protocol.
Arm/Group | Adolescents | Older Children | Young and Very Young Children
Serious Adverse Events (participants affected / at risk) | 0/21 | 1/28 | 0/17
Other Adverse Events (participants affected / at risk) | 12/21 | 20/28 | 6/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adolescents (N=21) | Older Children (N=28) | Young and Very Young Children (N=17)
post-procedural hemorrhage (Surgical and medical procedures) | 0 | 1 | 0 — Post-procedural hemorrhage occurred 6 days following tonsillectomy. Outside the therapeutic range of the investigational product.
OTHER ADVERSE EVENTS (reported when occurring in more than 3.6% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Adolescents (N=21) | Older Children (N=28) | Young and Very Young Children (N=17)
Nausea (Gastrointestinal disorders) | 6 | 9 | 1
Vomiting (Gastrointestinal disorders) | 3 | 8 | 0
Dizziness (Nervous system disorders) | 3 | 3 | 0
Headache (Nervous system disorders) | 2 | 0 | 2
Infusion site irritation (General disorders) | 0 | 0 | 1
Vessel puncture site bruise (General disorders) | 0 | 0 | 1
Cardiac murmur (Investigations) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Enlarged uvula (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 1 | 0
Somnolence (Nervous system disorders) | 1 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0
Diplopia (Eye disorders) | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hot flush (Vascular disorders) | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Otitis media (Infections and infestations) | 1 | 0 | 0
Otitis media viral (Infections and infestations) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Tremor (Nervous system disorders) | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
Another opioid may been given according to medical judgment/standard of care if the participant had persistent intolerable pain 2 hours or more after administration of tapentadol oral solution despite having received a non-opioid analgesic.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor reserves the right to review any publication pertaining to the trial before it is submitted for publication. Neither party has the right to prohibit publication unless publication can be shown to affect possible patent rights.